CLINICAL TRIAL: NCT05493397
Title: A Feasibility Study to Investigate the Accuracy and Viability of Ultrasound in Detecting Impairments of Vocal Fold Mobility in People With Neurological Disease
Brief Title: Ultrasound to Detect Vocal Fold Movement in Neurological Disease
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 146531
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Neurological Disorder; Ultrasound; Vocal Fold Movement
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the accuracy and viability of transcutaneous laryngeal ultrasound (US) in detecting impairments of vocal fold movement in people with neurological disorders.

The accuracy and viability of laryngeal US compared with reference standard fibreoptic nasendoscopic examination (FNE) will be evaluated. The study also includes measurements of clinician reliability in US image acquisition and interpretation, and assess the acceptability of US assessment to people with neurological disorders. Data will be used to assess the ability of US to detect other laryngeal pathology, and to calculate the sample size required for a validation study.

DETAILED DESCRIPTION:
The availability of cheaper and more portable ultrasound (US) machines has resulted in the extension of the use of US beyond the radiology department into diverse clinical areas. In particular, the Covid-19 pandemic has intensified interest in US as an alternative tool to use within the Speech and Language Therapy (SLT) profession to assess swallowing and airway disorders as access to routine assessment tools such as fibreoptic endoscopic examination (FNE) was restricted to its due aerosol-generating properties (Bolton et al., 2020).

The use of US by allied health professionals, such as Speech and Language Therapists (SLTs), is driven by National Institute for Health and Care Excellence (NICE) guidance and government policy (The Royal College of Radiologists, 2017) whereby the range of applications and locations where US can be used makes it impractical to deliver this imaging using radiologists or sonographers alone.

The application of laryngeal US is not new within the medical profession and there is considerable mounting evidence to support both the diagnostic ability and feasibility of laryngeal US for diagnosing impairments of vocal fold movement. Laryngeal US has been found to have both high sensitivity and specificity in diagnosing disorders of vocal fold movement in the post-surgical (specifically thyroid) population. Findings of a recent rapid review exploring the utility of laryngeal US for the assessment of vocal fold function revealed a sensitivity and specificity of 100% to detect normal versus disordered vocal fold function with a linear probe with range frequencies (e.g.6-13Hz) (Allen et al., 2020). To date, there are no studies exploring use of laryngeal US in assessing vocal fold movement in neurological conditions, despite the prominence of vocal fold impairments in this patient group.

In addition to increased accuracy, laryngeal US has many other advantages as an assessment and monitoring tool. Arguably, the greatest advantage of laryngeal US over FNE is its bedside accessibility and potential avoidance of intrusive procedures. This is particularly paramount in patients that require multiple invasive procedures, for example, combined FNE and non-invasive ventilation, cough augmentation, suction, nasogastric tube feeding and high flow oxygen therapy. Furthermore, if evaluation by laryngeal US was led by SLT, it would not require patient transport to Ear, Nose & Throat (ENT) clinics or presence of an ENT consultant at bedside; potentially expediting access to diagnosis of vocal fold function impairments and reducing cost.

A trained SLT could utilise US to identify presence or absence of vocal fold function impairment in patients with neurological disease. Primary examples are cases where vocal fold impairment is a known or anticipated symptom of the underlying neurological condition (such as brainstem stroke, multiple system atrophy and/or neuromuscular conditions such as Charot Marie Tooth disease). In these cases, the SLT could assess using laryngeal US to ascertain a vocal fold diagnosis to inform timely management or treatment plan. In cases where intrusive respiratory interventions may provoke issues with vocal fold movement (such as cough augmentation) the SLT can provide non-invasive 'real-time' monitored laryngeal US assessment which will directly influence combined SLT and physiotherapy management in patients with combined bulbar and respiratory disease. They could also use US to inform the relative urgency of subsequent ENT opinion. This is particularly pertinent at NHNN where there is no on-site access to ENT.

This research project is designed to improve the care pathway for patients with suspected vocal fold mobility impairment secondary to neurological disease. The current standard of practice for patients with suspected impairment of vocal fold mobility at our tertiary neurological centre is referral for routine assessment by an ENT doctor. The timescale from referral to assessment can be up to 12 weeks. FNE is an intrusive procedure requiring placement of a flexible scope into the throat via the nose. This can be uncomfortable for patients and, in some cases, contraindicated (Langmore, 2001). The clinical cost of an ENT-led nasendoscopy is £645. The procedure also requires pre- and post- assessment time and expertise for decontamination of the nasendoscope. Whereas, the cost of the US, led by and SLT is £62. The decontamination process is quick (using a simple wipe) and therefore more cost effective. Laryngeal US examination can be performed by an SLT within 48 hours of referral, leading to more timely assessment and intervention. Furthermore, preliminary findings from our patient advisory group indicate that US is a more comfortable and tolerable assessment. The outcomes of this study has the potential to influence clinical pathways at our tertiary centre to provide a service that is rapid, non-intrusive and cost-effective in the assessment for early diagnosis and management of vocal fold impairment.

This is a prospective cross-sectional mixed-methods study of consecutive patients referred from our tertiary neurological centre to ENT services for an assessment of their vocal fold mobility.

The study is to be conducted at a single-site, specialist tertiary centre, specialising in the diagnosis, assessment, and management of neurological disorders. It will adopt a cross-sectional design and aim to capture consecutive in- and out-patients with suspected vocal fold movement impairment referred to ENT for vocal fold assessment over the course of 12 months.

The anticipated sample size is n=50 patients.

Each research participant will be assessed once. The assessment will include the following (in order):

1. Invitation to participate which will include a patient information leaflet.
2. Signed consent.
3. TWO assessments, one of which is part of routine clinical care. These assessments are FNE and ii) Laryngeal US. FNE will be performed either by an ENT consultant or experienced SLT. A small, flexible camera is passed into the nose to view the throat. This assessment is part of routine clinical care (and is the current gold-standard for assessment for vocal fold movement. Laryngeal US uses a hand-held probe on the skin of the neck to assess the throat from the outside. Lubricating gel is used to improve contact between the skin and the probe.

   Each assessment will take less then 10 minutes to perform.
4. Participant survey. Each participant will be asked to complete a short (5-item) questionnaire to capture their experiences of undergoing each assessment.

As per usual clinical care - participants will receive a diagnosis from the ENT consultant based on the images from the FNE. They will be offered the opportunity to be contacted about the findings of the research study once data analysis is complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients under in-patient our out-patient Speech and Language Therapy care at primary study site.
* Patients with a neurological condition who have a suspected impairment of vocal fold movement due to diagnosis of dysphonia, breathing difficulties and/or impaired cough as determined by their lead Speech and Language Therapist.
* Over 18 years old
* Has undergone/will undergo nasendoscopy as part of their standard clinical care.

Exclusion Criteria:

* Patients who cannot be supported to demonstrate capacity to consent.
* Any patient that automatically meets the clinical exclusion criteria for FNE; e.g. epistaxis risk, facial fracture, patient distress.
* Patients who do not have sufficient command of English to consent in this study will also be excluded from the study due to limited resources for advocacy services. Participants will require sufficient English language skills to participate in the patient questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with neurological impairment due to be referred to Ear, Nose and Throat (ENT)services with suspected impairment of vocal fold function.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of transcutaneous laryngeal US in the diagnosis of vocal fold movement impairment in patients with neurological disease. | 12 months
  Each participant with be assessed using i) laryngeal ultrasound (US) and ii) fibreoptic nasendoscopic examination (FNE). One ENT or SLT will pass an FNE to assess vocal fold function. Images will be interpreted by an ENT consultant blinded to the outcomes of the laryngeal US. Two blinded SLTs will capture and interpret laryngeal US images. Each SLT will be blinded to the outcomes of i) the FNE assessment and ii) their SLT peer US assessment. Vocal fold movement will be assessed using a three-point scale (0 - normal movement, 1- impaired movement, 2- no movement).
  Descriptive and inferential statistics will be used to establish the sensitivity and specificity of laryngeal US in detecting an impairment of vocal fold movement impairment. A consensus agreement between the two blinded SLTs will be used to calculate the sensitivity and specificity.
Technical and environmental viability of laryngeal US in patients with neurological disease. | 12 months
  Image acquisition scored on a binary scale (possible/not possible). Any technical or environmental factors preventing US image acquisition will be captured on a pre-determined spread sheet.

SECONDARY OUTCOMES:
Reliability of assessors in capturing and interpreting laryngeal US images for the purpose of vocal fold movement assessment in patients with neurological disease. | 15 months
  Inter-rater reliability of the SLT US assessors will be calculated using kappa statistic.
Acceptability of transcutaneous laryngeal US to patients with neurological disease. | 15 months
  Each patient will be asked to complete a short survey about their experience of laryngeal US assessment. Quantitative data will be analysed descriptively. Qualitative data will be analysed using thematic analysis.
Diagnostic accuracy and feasibility of laryngeal US between patients of different neurological disease groups | 15 months
  Sub-group analysis will be used to explore the accuracy and feasibility of laryngeal US according to neurological diagnosis.
Ability of US to detect other laryngeal pathology in patients with neurological disease. | 24 months
  Where additional laryngeal pathology was diagnosed on FNE, retrospective analysis of these images will be conducted alongside US images to generate hypothesis relating to the ability of US to detect other laryngeal pathology in this patient group. Findings will be descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Allen, Principal Investigator — University College London Hospitals
Locations (1):
- University College London Hospitals, London, United Kingdom

REFERENCES:
- [Background] Bolton L, Mills C, Wallace S, Brady MC; Royal College of Speech and Language Therapists (RCSLT) COVID-19 Advisory Group. Aerosol generating procedures, dysphagia assessment and COVID-19: A rapid review. Int J Lang Commun Disord. 2020 Jul;55(4):629-636. doi: 10.1111/1460-6984.12544. Epub 2020 Jun 1. No abstract available. PMID 32478950
- [Background] Allen J, Clunie G, Slinger C et al. Utility of ultrasound in the assessment of swallowing and laryngeal function: A rapid review and critical appraisal of the literature. International Journal of Language and Communication Disorders 2021 56 (1): 174-204.
- [Background] Langmore SE. Endoscopic Evaluation and Treatment of Swallowing Disorders. 2001. New York: Thieme Publishers